CLINICAL TRIAL: NCT06904053
Title: Metagenomics Next-Generation Sequencing Approach to Detect Microbial DNA/RNA Overtime in Individuals Undergoing Hematopoietic Stem Cell Transplant
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10001923; 001923-CC
Record Dates: First submitted 2025-03-29; First posted 2025-04-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11-19

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Microbial DNA/RNA; Hematopoietic stem cell transplant (HSCT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All HSCT patients: Male or female, aged 3 years or older.

SUMMARY:
Infections are a major cause of morbidity and mortality in patients undergoing hematopoietic stem cell transplant (HSCT). The purpose of this study is to evaluate if metagenomic next-generation sequencing (mNGS) can detect microbial signatures in people undergoing HSCT, and if microbial identification can be correlated with clinical features of infection (e.g., fever). Participants undergoing HSCT as part of other studies at the NIH Clinical Center (CC) will provide blood before the transplant and through 6 months after. Total nucleic acid will be extracted from plasma and subjected to mNGS.

The primary objective of this study is to investigate if by using plasma and an mNGS approach, we can detect bacterial, fungal, protozoan, or viral DNA/RNA over time, in immunocompromised patients undergoing transplantation.

Secondary objectives are to: (1) To correlate microbial identification with episodes of fever or clinical suspicion of infection; and to (2) correlate change in microbial signatures in patients with suspected immune reconstitution inflammatory syndrome.

The study is conducted at the NIH Clinical Center. Participants, aged 3 years and older, on other research studies at the NIH CC who are undergoing HSCT are invited to take part of this study. Expected participation is up to six months.

DETAILED DESCRIPTION:
Study Description:

Infections are a major cause of morbidity and mortality in patients undergoing hematopoietic stem cell transplant (HSCT). The purpose of this study is to evaluate if metagenomic next-generation sequencing (mNGS) can detect microbial signatures in people undergoing HSCT, and if microbial identification can be correlated with clinical features of infection (e.g., fever).

Participants undergoing HSCT as part of other studies at the NIH Clinical Center (CC) will provide blood before the transplant and through 6 months after. Total nucleic acid will be extracted from plasma and subjected to mNGS.

Objectives:

Primary:

To investigate if by using plasma and an mNGS approach, we can detect bacterial, fungal, protozoan, or viral DNA/RNA over time, in immunocompromised patients undergoing transplantation.

Secondary:

1. To correlate microbial identification with episodes of fever or clinical suspicion of infection.
2. To correlate change in microbial signatures in patients with suspected immune reconstitution inflammatory syndrome.

Endpoints:

Primary:

Comparison of mNGS results to routine clinical test results (microbiology and/or pathology)

Secondary:

1. Calculation of frequencies of different microbial identifications as it relates to the development of fever or microbiologically/clinically defined infection.
2. Changes in different microbial signatures over time

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study; an individual must meet all the following criteria:

1. Male or female, aged 3 years or older.
2. Co-enrolled on another study at the NIH CC, under which they will undergo HSCT.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual with any condition that, in the opinion of the investigator, contraindicates participation in this study, will be excluded.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged 3 years and older on other research studies at the NIH CC who are undergoing HSCT as part of that study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Any positive clinical results for each of 5 pathogen categories | Six months
  Research blood draw at screening, during fever episodes and at follow up days 30, 100 and 180 (+/- 7 days).

CONTACTS AND LOCATIONS:
Overall Officials: Sanchita Das, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001923-CC.html